CLINICAL TRIAL: NCT01434446
Title: The Effect of Sound Stimulation on Hearing Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Earlogic Korea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEK 08252011
Record Dates: First submitted 2011-09-09; First posted 2011-09-15 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

INTERVENTIONS:
Behavioral: Sound stimulation — Listening to sound stimuli at the lowest audible level.

SUMMARY:
In the late 1990s, researchers discovered that acoustic stimuli slow progressive sensorineural hearing loss and exposure to a moderately augmented acoustic environment can delay the loss of auditory function. In addition, prolonged exposure to an augmented acoustic environment could improve age-related auditory changes. These ameliorative effects were shown in several types of mouse strains, as long as the acoustic environment was provided prior to the occurrence of severe hearing loss.

In addition to delaying progressive hearing loss, acoustic stimuli could also protect hearing ability against damage by traumatic noise. In particular, a method called forward sound conditioning (i.e., prior exposure to moderate levels of sound) has been shown to reduce noise-induced hearing impairment in a number of mammalian species, including humans.

Interestingly, recent report has suggested that low-level sound conditioning also reduces free radical-induced damage to hair cells, increases antioxidant enzyme activity, and reduces Cox-2 expression in cochlea, and can enhance cochlear sensitivity. Specifically, increased cochlear sensitivity was observed when distortion product otoacoustic emissions (DPOAEs) and compound action potentials (CAPs) were measured.

In addition to forward sound conditioning, backward sound conditioning (i.e., the use of acoustic stimuli after exposure to a traumatic noise) has been shown to protect hearing ability against acoustic trauma and to prevent the cortical map reorganization induced by traumatic noise.

In this study, the investigators examine the effect of sound stimulation on hearing ability in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age between 20 and 70 years
* Subjects should be able to use an mp3 player

Exclusion Criteria:

* Hearing loss more than 70 dB HL at any frequency
* More than 10 dB of air-bone gaps at more than 3 frequencies in pure-tone audiometry
* Ear infections, chronic middle ear disease or any abnormality of the ear canal or ear drum
* Temporary hearing loss
* Hearing aid user
* Pregnant females

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Changes of pure-tone hearing thresholds after sound stimulation | 2~6 months
  Pure-tone hearing thresholds of the baseline and the final point (after 2~6 months)will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Eunyee Kwak, Ph.D., Principal Investigator — Earlogic Auditory Research Institute
Locations (1):
- Earlogic Auditory Research Institute, Seoul, South Korea